CLINICAL TRIAL: NCT04632680
Title: ECG-I Targeted Ablation for Persistent AF
Acronym: TARGET-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 218367-2
Record Dates: First submitted 2020-11-11; First posted 2020-11-17 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation ECG-I Mapping Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- PVI followed by targeting of drivers (Experimental): Patients will undergo intra-procedural mapping using the ECG-I. The pulmonary veins will be isolated. Drivers will then be targeted as guided by the ECG-I system aiming for termination of AF.
  Interventions: Device: PVI followed by targeting of drivers

INTERVENTIONS:
Device: PVI followed by targeting of drivers — Patients will undergo intraprocedural ECG-I mapping. The pulmonary veins will be isolated followed by targeting of drivers aiming to terminate AF.

SUMMARY:
Atrial fibrillation (AF) is an irregular heart rhythm associated with significant morbidity and mortality. Catheter ablation is an established treatment where catheters are inserted through a vein in the leg into the left atrium of the heart to deliver lines of scar to disrupt the tissue causing and maintaining AF.

The ECG-I is a system which involves wearing a jacket with many ECG electrodes to record electrical activity from the surface of the body. A CT scan then shows where these electrodes are relative to the atria, and computer modelling is used to reconstruct the movements of electricity on the surface of the heart and therefore identifying where the drivers (tissue causing and maintaining AF) are located.

Success rates for persistent atrial fibrillation lie in the region of 30-60% due to the location of drivers (tissue causing and maintaining AF) varying per patient. Locating and treating these drivers is very challenging.

We intend to enrol 40 patients with persistent AF and perform atrial mapping using the ECG-I system. We will perform pulmonary vein isolation and perform atrial mapping to identify the location of these drivers and then to ablate them. We will study the effects of performing ablation upon these drivers using the ECG-I.

DETAILED DESCRIPTION:
Atrial Fibrillation (AF) is the commonest heart rhythm disturbance and is associated with significant morbidity and mortality. Catheter ablation (CA) is a procedure where catheters (leads) are passed into the heart and energy is used to disrupt and isolate (by freezing or cauterising) heart tissue causing AF. CA is an established therapy for AF. Success rates for CA for paroxysmal AF lies in the region of 70% or better. However, success rates for persistent AF is much lower and estimates lie in the region of 30-60%.

Current CA protocols for AF centre on isolating the pulmonary veins (the pulmonary veins drain into the left atrium) which have been proven to trigger AF. Pulmonary Vein Isolation (PVI) ablation alone seems sufficient to remove the trigger for the vast majority of patients with paroxysmal AF. However, in patients with persistent AF it is common for AF to continue after the pulmonary veins have been electrically isolated.

The difference in success rates between the paroxysmal and persistent form of AF is thought to be due to changes within the heart atria after AF has been established for some time. In persistent AF the atria dilate and remodel structurally and electrically, and therefore the maintenance of persistent AF differs from paroxysmal AF.

Persistent AF is thought to be maintained by focal sources, whether rotors or sites of radial activation. Currently, targeting other sites within the atria in addition to PVI such as fractionated electrograms (areas of electrical activity) are thought to be imprecise and require extensive ablation. Often AF will persist despite targeting additional sites within the atria.

Currently clinical characteristics of patients or structural imaging have limited accuracy in selecting patients likely to benefit from CA. Mapping studies have shown that patients with persistent AF who have higher frequency signals near the pulmonary veins than being distributed in the left atrial body are more likely to terminate to sinus rhythm (normal heart rhythm) with PVI alone and to maintain sinus rhythm.

Studies have suggested that patients undergoing standard PVI ablation procedures for persistent AF who have coincidental interruption of drivers have a far better long term outcome. This suggests that the characteristics of atrial heart tissue and electrical activation patterns maintaining AF are likely to determine the response to ablation therefore it may be possible to determine more directly and accurately the likelihood of success by performing non-invasive mapping of the atria using the ECG-I.

ECG-I is able to localise the drivers of AF and one of the objectives is to study the electrical characteristics of the tissue. ECG-I is currently being used in research into AF. A recently published a study using ECG-I to identify targets of ablation in 103 patients. They suggested that using ECG-I may improve CA success rates and reduces the procedure time and amount of ablation. The prospective multicentre AFACART study had similar findings.

We intend to enrol 40 patients who will undergo Atrial Mapping with ECG-I during catheter ablation. After isolation of the pulmonary veins patients drivers will be targeted guided by the system.

ELIGIBILITY:
Inclusion Criteria:

* Persistent AF (i.e. episodes of AF that are continuous for > 1 week)
* Willing for ablation.
* Age between 18 to 80.

Exclusion Criteria:

* Duration of continuous persistent AF > 2 years
* Left atrial diameter > 5 cm
* Severe left ventricular impairment (EF < 40%)
* New York Heart Association class 3 or 4 heart failure
* Known hypertrophic cardiomyopathy, cardiac sarcoid or Arrhythmogenic cardiomyopathy.
* Known inherited arrhythmia such as Brugada or long QT syndromes
* Valvular disease that is more than moderate
* History of valve replacement (metallic or tissue)
* History of congenital heart disease (other than patent foramen ovale)
* Previous left atrial ablation (percutaneous or surgical)
* Cardiac surgery or percutaneous coronary intervention within the last 3 months.
* Myocardial infarction or unstable angina within the last 3 months.
* Unwillingness for ablation
* Unwillingness to be involved in study
* Suspected reversible cause of AF
* Any other contraindication to catheter ablation
* Age < 18 yrs or > 80 years
* Pregnancy
* Morbid obesity (defined as body mass index >40)
* Any other medical problem likely to cause death within the next 18 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Number of participants free from atrial arrhythmia (including AF and atrial tachycardia) at 12 months | 12 months
  Number of participants free from atrial arrhythmia (including AF and atrial tachycardia) at 12 months

SECONDARY OUTCOMES:
Number of participants free from Atrial Fibrillation at 12 months | 12 months
  Number of participants free from Atrial Fibrillation at 12 months.
Termination of AF with PVI followed by ECGI guided driver ablation | During Catheter Ablation Procedure
  Rates of termination of AF intra-procedurally during ablation
Composite end point including rates of AF termination and cycle length slowing with PVI followed by ECGI guided driver ablation | During Catheter Ablation Procedure
  Rates of reaching composite end point (either termination of AF or cycle length slowing) intra-procedurally during ablation

CONTACTS AND LOCATIONS:
Overall Officials: Ross Hunter, Principal Investigator — Barts Heart Centre
Locations (1):
- Barts Heart Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided